CLINICAL TRIAL: NCT07128680
Title: A Randomized Study of Nivolumab and Ipilimumab With and Without EXL01 in First-Line Treatment of Metastatic Renal Cell Carcinoma (mRCC)
Brief Title: Immunotherapy (Nivolumab and Ipilimumab) With and Without a Live Biotherapeutic Product (EXL01) for the Treatment of Metastatic Renal Cell Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25160; NCI-2025-05679 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25160 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-08-14; First posted 2025-08-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Advanced Clear Cell Renal Cell Carcinoma; Advanced Sarcomatoid Renal Cell Carcinoma; Metastatic Clear Cell Renal Cell Carcinoma; Metastatic Sarcomatoid Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Carcinoma, Renal Cell | interventions — Specimen Handling; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (nivolumab, ipilimumab, EXL01) (Experimental): CYCLES 1-4: Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1 of each cycle and receive EXL01 PO QD on days 1-21 of each cycle. Cycles repeat every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  CYCLES 5+: Patients continue receiving nivolumab IV over 30 minutes on day 1 of each cycle and EXL01 PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Patients also undergo CT and collection of blood samples throughout the study. Patients may undergo MRI at screening and may undergo bone scan as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Dietary Supplement: Faecalibacterium prausnitzii-containing Bacterial Strain Formulation EXL01; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab
- Arm B (nivolumab, ipilimumab) (Active Comparator): CYCLES 1-4: Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  CYCLES 5+: Patients continue receiving nivolumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Patients also undergo CT and collection of blood samples throughout the study. Patients may undergo MRI at screening and may undergo bone scan as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Dietary Supplement: Faecalibacterium prausnitzii-containing Bacterial Strain Formulation EXL01 — Given PO
  Other Names: EXL 01; EXL-01; EXL01; F. prausnitzii-containing Bacterial Strain Formulation EXL01
  Arms: Arm A (nivolumab, ipilimumab, EXL01)
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This phase I trial tests the safety and effectiveness of nivolumab and ipilimumab with and without EXL01 for the treatment of renal cell cancer that has spread from where it first started (primary site) to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. EXL01 is a live biotherapeutic product containing a strain of bacteria called Faecalibacterium prausnitzii. It may enhance a patient's response to treatment with immune checkpoint inhibitors like nivolumab and ipilimumab by altering the composition of the bacteria in the gut. Adding EXL01 to treatment with nivolumab and ipilimumab may be safe and more effective than giving nivolumab and ipilimumab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effects of Faecalibacterium prausnitzii-containing bacterial strain formulation EXL01 (EXL01) (in combination with nivolumab/ipilimumab) on systemic immunomodulation in patients with mRCC.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of EXL01 (in combination with nivolumab/ipilimumab) in the treatment of patients with mRCC.

II. To evaluate the effect of EXL01 on the clinical efficacy of nivolumab/ipilimumab.

EXPLORATORY OBJECTIVES:

I. To determine the effect of EXL01 on gut microbiome diversity and function. II. To determine the effect of EXL01 on systemic immunodulation.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A:

CYCLES 1-4: Patients receive nivolumab intravenously (IV) over 30 minutes and ipilimumab IV over 30 minutes on day 1 of each cycle and receive EXL01 orally (PO) once daily (QD) on days 1-21 of each cycle. Cycles repeat every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

CYCLES 5+: Patients continue receiving nivolumab IV over 30 minutes on day 1 of each cycle and EXL01 PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients also undergo computed tomography (CT) and collection of blood samples throughout the study. Patients may undergo magnetic resonance imaging (MRI) at screening and may undergo bone scan as clinically indicated.

ARM B:

CYCLES 1-4: Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

CYCLES 5+: Patients continue receiving nivolumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients also undergo CT and collection of blood samples throughout the study. Patients may undergo MRI at screening and may undergo bone scan as clinically indicated.

After completion of study treatment, patients are followed up within 30 days then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: ≥ 18 years at time of signing informed consent
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Life expectancy > 3 months
* Histologically confirmed renal cell carcinoma with clear cell renal cell carcinoma component with or without sarcomatoid component
* Advanced (not amenable to curative surgery or radiation therapy) or metastatic (American Joint Committee on Cancer [AJCC] stage IV) renal cell carcinoma with any disease risk disease by International Metastatic RCC Database Consortium (IMDC) criteria (good-, intermediate- or poor-risk)
* No prior systemic therapy for RCC with the following exception:

  * One prior adjuvant or neoadjuvant therapy for completely resectable RCC if recurrence occurred at least 6 months after the last dose of adjuvant or neoadjuvant therapy, provided that the patient has fully recovered from acute toxic effects to prior anti-cancer therapy
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Absolute neutrophil count (ANC) ≥ 1,000/mm^3

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement
* Platelets ≥ 100,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement
* Hemoglobin ≥ 9g/dL

  * NOTE: Red blood cell transfusions are not permitted within 14 days of hemoglobin assessment unless cytopenia is secondary to disease involvement
* Total bilirubin ≤ 1.5 X upper limit of normal (ULN) (except for subjects with Gilbert Syndrome, who may have total bilirubin up to 3.0 mg/dL)
* Aspartate aminotransferase (AST) ≤ 3.0 x ULN
* Alanine aminotransferase (ALT) ≤ x ULN
* Creatinine clearance of ≥ 30 mL/min per 24-hour urine test or the Cockcroft-Gault formula or serum creatinine < 1.5 x upper limit of normal (ULN)
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin (PT) ≤ 1.5 x ULN
* If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN
* If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants
* If seropositive for HIV, hepatitis C virus (HCV) or hepatitis B virus (HBV), nucleic acid quantitation must be performed. Viral load must be undetectable. HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Meets other institutional and federal requirements for infectious disease titer requirements

  * Note infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test within 72 hours of study start

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 5 months after the last dose of nivolumab or ipilimumab for women with childbearing potential, and 5 months after the last dose of nivolumab or ipilimumab for men. For EXL01, female participants should continue contraception for 30 days after the last dose
* Female subjects of childbearing potential must not be pregnant at screening. Female subjects are considered to be of childbearing potential unless one of the following criteria is met: documented permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating [FSH] level > 40 mIU/mL to confirm menopause).

  * Note: Documentation may include review of medical records, medical examinations, or medical history interview by study site

Exclusion Criteria:

* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Current use, or intent to use probiotics, prebiotics, bacterial fortified foods and other natural supplements ≤ 2 week prior to treatment initiation and during the period of treatment
* Any botanical preparation (e.g. herbal supplements or traditional Chinese medicines) intended to treat the disease under study or provide supportive care
* Fecal microbiota transplant within 3 months prior to screening

  * Note: Patients must have recovered adequately from the toxicity and/or complications from the treatment prior to starting study intervention
* Patients requiring chronic antibiotic therapy at the time of study enrollment
* Unstable cardiac disease as defined by one of the following:

  * Cardiac events such as myocardial infarction (MI) within the past 6 months
  * NYHA (New York Heart Association) heart failure class III-IV
  * Uncontrolled atrial fibrillation or hypertension
* Active interstitial lung disease (ILD)/pneumonitis or history of ILD/pneumonitis requiring treatment with systemic steroids
* Known medical condition (e.g., a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results
* Receipt of any type of cytotoxic, biologic, or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment
* Radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Patients must have recovered adequately from the toxicity and/or complications from the treatment prior to starting study intervention
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks prior to first dose of study treatment after radiotherapy or at least 4 weeks prior to first dose of study treatment after major surgery (e.g., removal or biopsy of brain metastasis). Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment
* Administration of a live, attenuated vaccine within 30 days before first dose of study treatment
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days before first dose of study treatment

    * Note: Inhaled, intranasal, intra-articular, or topical steroids are permitted. Adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent are permitted. Transient short-term use of systemic corticosteroids for allergic conditions (e.g., contrast allergy) is also allowed
  * History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* Active inflammatory intestinal disease (Crohn disease, Hemorrhagic recto-colitis, coeliac disease) or any serious chronic intestinal disease with uncontrolled diarrhea
* Known positive test for tuberculosis infection where there is clinical or radiographic evidence of active mycobacterial infection
* Major surgery within 28 days (4 weeks) prior to first dose of study treatment

  * Note: Participants who had surgery > 4 weeks prior to screening must have recovered adequately from any toxicity and/or complications from the surgery or trauma prior to starting study intervention
* Malabsorption syndrome
* Uncompensated/symptomatic hypothyroidism
* Moderate to severe hepatic impairment (Child-Pugh B or C)
* Requirement for hemodialysis or peritoneal dialysis
* History of solid organ or allogenic stem cell transplant
* Other clinically significant disorders that would preclude safe study participation.

  * Any active, known, or suspected autoimmune disease will be excluded, with the following exceptions:

    * Type 1 diabetes mellitus.
    * Hypothyroidism only requiring hormone replacement.
    * Skin disorders (e.g., vitiligo, psoriasis, or alopecia) not requiring systemic treatment.
    * Conditions not expected to recur in the absence of an external trigger
* Gastrointestinal (GI) obstruction, poor oral intake, or difficulty in taking oral medication or difficulties in swallowing; nasogastric tubes are not permitted or unwillingness or inability to receive IV administration
* Known history or newly diagnosed GI parasitic infection within 3 months prior to screening. Patients must have recovered adequately from the toxicity and/or complications from the treatment prior to starting study intervention
* Previously identified allergy or hypersensitivity to components of the study treatment formulations or history of severe infusion-related reactions to monoclonal antibodies. Subjects with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption are also excluded
* A patient with a known serious hypersensitivity to any component of the drug formulation for EXL01, or any other live biotherapeutic product (LBP), should not receive EXL01
* Hypersensitivity to soy products
* Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to first dose of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-06-02 (Estimated); Study Completion 2027-06-02 (Estimated)

PRIMARY OUTCOMES:
Change in plasma IFNγ | At baseline and week 13
  IFNγ plasma concentration will be analyzed using a 2-sample t-test if normality assumptions are met; otherwise, the Wilcoxon rank sum test will be applied.

SECONDARY OUTCOMES:
Incidence of grade ≥ 3 adverse events (AEs) | Up to 30 days after last dose of treatment
  The safety evaluation will be based on all patients that received at least one dose of the drug and will include AEs, serious AEs, and changes from baseline in laboratory evaluations, vital signs, and physical examinations. Summaries will be provided overall and by treatment group. The number and percentage of subjects reporting treatment-emergent AEs (TEAE) will be summarized overall and by the worst Common Terminology Criteria for Adverse Events grade. Similarly, the number and percentage of subjects reporting TEAEs considered related to each study drug will be summarized.
Best overall response | Up to 2 years
  Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria. The association between treatment arm and overall response as per RECIST criteria (response observed versus not observed) will be examined using Fisher's exact test.
Duration of response | From first documented complete response or partial response until disease progression or death, assessed up to 2 years
Progression free survival | From start of treatment to time of progressive disease or death, assessed up to 2 years
  The difference in progression free survival across the two groups will be explored graphically using Kaplan-Meier survival plots. Median progression-free survival time for each of the two arms will be reported and Cox Proportional Hazards model will be used to estimate the hazard ratio and its confidence interval.
Overall survival | From start of treatment to death from any cause, assessed up to 2 years
  The difference in overall survival across the two groups will be explored graphically using Kaplan-Meier survival plots. Median overall survival time for each of the two arms will be reported. A Cox Proportional Hazards model will be used to estimate the hazard ratio and its 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Sumanta K Pal, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Medical Center, Irvine, California